CLINICAL TRIAL: NCT05602961
Title: A Phase I/II Partially Randomized, Active-controlled Observer-blind, Dose-selection, Safety and Immunogenicity Study of GLB-COV2-043, an mRNA Vaccine Candidate Against SARS-CoV-2, Administered as a Single-vaccination Booster to Previously Vaccinated Adults
Brief Title: A Phase I/II Study of GLB-COV2-043 as a COVID-19 Vaccine Booster
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: to prioritize other programs.
Sponsor: GreenLight Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GLB-003
Record Dates: First submitted 2022-10-28; First posted 2022-11-02 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (includes GLB-COV2-043 15 μg) (Experimental): 12 eligible adult participants will be randomized to 15 ug of GLB-COV2-043 or to 30 ug of BNT162b2/COMIRNATY®, active control with a 5:1 allocation ratio.
  Interventions: Drug: GLB-COV2-043; Drug: BNT162b2/COMIRNATY®
- Cohort 2 (includes GLB-COV2-043 30 μg) (Experimental): 12 eligible adult participants will be randomized to 30 ug of GLB-COV2-043 or to 30 ug of BNT162b2/COMIRNATY®, active control with a 5:1 allocation ratio.
  Interventions: Drug: GLB-COV2-043; Drug: BNT162b2/COMIRNATY®
- Cohort 3 (includes GLB-COV2-043 60 μg) (Experimental): 12 eligible adult participants will be randomized to 60 ug of GLB-COV2-043 or to 30 ug of BNT162b2/COMIRNATY®, active control with a 5:1 allocation ratio.
  Interventions: Drug: GLB-COV2-043; Drug: BNT162b2/COMIRNATY®
- Cohort 4 (includes GLB-COV2-043 90 μg) (Experimental): 12 eligible adult participants will be randomized to 90 ug of GLB-COV2-043 or to 30 ug of BNT162b2/COMIRNATY®, active control with a 5:1 allocation ratio.
  Interventions: Drug: GLB-COV2-043; Drug: BNT162b2/COMIRNATY®

INTERVENTIONS:
Drug: GLB-COV2-043 — COVID-19 vaccine, administered as a booster
Drug: BNT162b2/COMIRNATY® — active control

SUMMARY:
The scope of this Phase I/II study is to determine whether GLB-COV2-043 is a promising booster vaccine candidate component for adult participants who have received the 2-dose priming course of the mRNA BNT162b2 vaccine against COVID-19, or the 2-dose priming course and a third BNT162b2 injection (i.e., as a "booster"), and, if so, to select the booster dose for further evaluation and potential development.

ELIGIBILITY:
Inclusion Criteria

1. The participant is ≥ 18 years of age (yoa) at the time of signing the informed consent form.
2. The participant provides documentation of completing the priming schedule, or the priming schedule and a third vaccination (i.e., a "booster"), with the mRNA BNT162b2 vaccine against SARS-CoV-2 at least 3 months before randomization.
3. The participant is willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study.
4. In the judgement of the investigator or designee, the participant has understood the information provided and the potential impact and/or risks linked to study vaccine administration and to participation in the study; written informed consent will be obtained from the participant before any study-related procedure is performed.
5. In the judgement of the investigator or designee, the participant is in good health as assessed by medical history, physical examination, and laboratory tests.
6. If a person of childbearing potential and sexually active, the participant is willing to commit to use an effective method of contraception from at least 1 week before randomization to 52 weeks after randomization.
7. If a person of childbearing potential, the participant is willing to undergo urine pregnancy tests as required by the protocol.

Exclusion Criteria

1. Medical conditions. The participant has:

   i. Current COVID-19 as determined by a positive SARS-CoV-2 RT-PCR at screening or a positive SARS-CoV-2 rapid antigen test at Visit 2.

   ii. History of SARS-CoV-2 infection or COVID-19 within 3 months before randomization, per volunteer self-report.

   iii. History of significant local or systemic hypersensitivity to vaccines, including mRNA vaccines or excipients (e.g., anaphylaxis, respiratory difficulties, angioedema, injection site necrosis, or ulceration) at any time.

   iv. History of splenectomy at any time. v. Ongoing or history of immunodeficiency or autoimmune disease at any time (not excluded: mild psoriasis that does not require ongoing systemic treatment).

   vi. Ongoing or history of myocarditis or pericarditis at any time vii. Ongoing or history of malignancy that, in the judgement of the investigator, has potential for recurrence (excluding basal cell carcinoma).

   viii. Ongoing or history of seizures requiring medication (not excluded: febrile seizures before the age of 5 or seizures secondary to alcohol withdrawal more than 3 years ago).

   ix. Ongoing suicidal thoughts or history of suicide attempt in the last 3 years.

   x. Ongoing or history of clinically significant substance or alcohol abuse in the last 3 years.

   xi. History of blood transfusion in the last 6 months. xii. Ongoing or history of bleeding disorder diagnosed by a healthcare provider (e.g., factor deficiency or coagulopathy).

   xiii. Ongoing or history of infections requiring antibiotic, antiviral or antifungal therapy in the last 1 month.

   xiv. Ongoing or history of any other clinically relevant medical condition, including serious psychiatric disorders, that in the judgement of the investigator or designee makes the participant unsuitable for participation in the study.
2. Vaccines. The participant has:

   i. Received a COVID-19 vaccine other than 2 or 3 doses of an authorized or approved mRNA COVID-19 vaccine.

   ii. Received only 1 dose of an authorized mRNA vaccine. iii. Received a fourth dose (i.e., more than one booster) of a COVID-19 vaccine.

   iv. Received any vaccine in the last 28 days or plans to receive any vaccine in the 6 months after the booster vaccine administration, with the exception of subunit influenza vaccines, which may be administered ≥ 7 days after study vaccine administration.
3. Medications. The participant has:

   i. Ongoing or history of use of immunosuppressive medications in the last 6 months.

   ii. Ongoing or history of use of systemic corticosteroids in the last 2 months (use of topical or inhaled steroids is permitted).

   iii. Ongoing or history of intake of any other medication that in the judgement of the investigator or designee makes the participant unsuitable for participation in the study.
4. The participant is lactating, pregnant or planning a pregnancy in the 12 months after randomization.
5. Laboratory tests. The participant has any of the following test results at screening:

   i. Positive test for HIV-1, HIV-2, hepatitis B, hepatitis C. ii. Haemoglobin ≤ 10.5 g/dl or ≤ 6.5 mmol/L in volunteers assigned female sex at birth; ≤ 11.0 g/dl or ≤ 6.8 mmol/L in volunteers assigned male sex at birth.

   iii. Leukocyte (WBC) count ≥ 12,000 cells/mm3 OR ≤ 3,000 cells/mm3 iv. Platelet count ≤ 125,000 cells/mm3 or ≤ 125 × 109 cells/L. v. Creatinine ≥ 1.1 × upper limit of normal (ULN). vi. Alanine transaminase (ALT) ≥ 1.25 × ULN.
6. The participant is enrolled in another interventional clinical trial or was enrolled in the last 3 months or plans to participate during this study (concurrent participation in an observational study not requiring blood or tissue sample collection is allowed).
7. In the judgement of the investigator or designee it is not in the best interest of the participant to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-21 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Safety, including reactogenicity | Day 0 to Day 28 post-vaccination
  * Proportion of participants experiencing severe (Grade ≥ 3) solicited treatment emergent AEs
  * Proportion of participants with severe (Grade ≥ 3) non-serious unsolicited treatment emergent AEs
  * Proportion of participants with serious unsolicited treatment emergent AEs (SAEs)
Immunogenicity- neutralizing antibody response | Day 0 to Day 28 post-vaccination
  Geometric mean titre (GMT) and geometric mean ratios (GMR) relative to baseline of neutralizing IgG antibodies against the spike (S) protein of the SARS-CoV-2 Wuhan strain

SECONDARY OUTCOMES:
Safety, including reactogenicity | Day 0 to Day 168 post-vaccination
  * Proportion of participants experiencing solicited treatment emergent AEs
  * Proportion of participants experiencing unsolicited treatment emergent AEs
  * Proportion of participants experiencing AEs of special interest (AESI), AEs requiring unscheduled medical attendance (MAAEs) or Serious AEs (SAEs)
Antibody-mediated immunogenicity titers (GMT) | baseline (Week 0) and 4, 24 and 52 weeks (7, 28, 168 and 365 days) post-vaccination
  Serum neutralizing IgG antibodies and binding IgG antibodies against the spike (S) protein of the original (wild) Wuhan strain, Omicron Variant of Concern (VoC), Delta VoC, Beta VoC, and Gamma VoC assessed as geometric mean titres (GMT), geometric mean ratio (GMR, fold increase from baseline) and percentage of sero-responders
Antibody-mediated immunogenicity fold-increase (GMR) | baseline (Week 0) and 4, 24 and 52 weeks (7, 28, 168 and 365 days) post-vaccination
  Serum neutralizing IgG antibodies and binding IgG antibodies against the spike (S) protein of the original (wild) Wuhan strain, Omicron Variant of Concern (VoC), Delta VoC, Beta VoC, and Gamma VoC assessed as geometric mean ratio (GMR, fold increase from baseline) and percentage of sero-responders
Antibody-mediated immunogenicity response rate | baseline (Week 0) and 4, 24 and 52 weeks (7, 28, 168 and 365 days) post-vaccination
  Serum neutralizing IgG antibodies and binding IgG antibodies against the spike (S) protein of the original (wild) Wuhan strain, Omicron Variant of Concern (VoC), Delta VoC, Beta VoC, and Gamma VoC assessed as percentage of sero-responders
Cell-mediated immunogenicity | 4 and 24 weeks (28 and 168 days) post-vaccination
  Intracellular cytokine staining (ICS) of antigen specific CD4+ and CD8+ T-cells against the original (wild) Wuhan strain, Omicron VoC and Delta VoC assessed as frequency of total antigen-specific CD4+ and CD8+ T-cells producing IFN-gamma, TNF-alpha or IL-2

CONTACTS AND LOCATIONS:
Overall Officials: Shelly Karuna, MD, MPH, Study Director — GreenLight Biosciences; Etienne Karita, MD, MSc, MSPH, Principal Investigator — Center for Family Health Research